CLINICAL TRIAL: NCT06607341
Title: Community Engagement ALliance Against Disparities - Washington District of Columbia (DC), Maryland, and Virginia (CEAL-DMV)
Brief Title: Community Engagement Alliance Against Disparities
Acronym: CEAL-DMV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Baltimore CONNECT (Unknown); Coaching Salud Holistica (Unknown); La Clinica del Pueblo (Unknown); Rivera Group (Unknown); The Medi Inc. (Unknown); Westat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IRB00338867; 6922-03-COVID-S017 (Other Grant/Funding Number: Westat Inc./NIH-NHLBI)
Record Dates: First submitted 2024-09-01; First posted 2024-09-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Diabetes; Pre-diabetes; Hypertension; Overweight and Obesity
Keywords: CEAL-DMV; Community Engagement Alliance; Diabetes; Hypertension; Pre-diabetes
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Hypertension; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized delayed control group with phased recruitment design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-level, community-digital health promotion intervention (Experimental): Participants will receive a multi-level, community-digital health promotion intervention.
  1. Community-level: Community Health Workers will assess needs of individuals including through a survey and facilitate access to the Medi digital resource platform.
  2. Individual level: CHW-delivered coaching on behavior-change goals and facilitation to services via the Medi platform. Participants will also receive tailored social media and in person reinforcements and cues to action based on goal attainment
  3. Social network level: Participants will receive tailored recommendations sent via social media on nearby parks, recreational facilities, faith-based ministries, and peer groups to support behavior change goals
  Interventions: Behavioral: Multi-level, community-digital health promotion intervention
- Delayed control intervention group (Active Comparator): At the individual level, participants will receive standardized 12-month text message (SMS) campaign. At the community-level, the investigators will equip community-based organization partners and community health workers with chronic disease educational content. Participants will also receive recommendations for health events and fairs locally.
  Interventions: Behavioral: Multi-level, community-digital health promotion intervention

INTERVENTIONS:
Behavioral: Multi-level, community-digital health promotion intervention — Community level activities:
  1. Capacity building for community-based organizations, and
  2. Community health workers will facilitate linkage to community resources, including health/social service access referrals and client social support.
  Individual level activities:
  1. Goal setting and self-monitoring,
  2. Tailored feedback,
  3. Personalized lifestyle coaching, health and social service referral support, and
  4. Digital access and digital health literacy skills building
  Social network:
  1. Social network-based activities, and
  2. Digital health literacy skills building

SUMMARY:
The Community Engagement Alliance against Disparities - Washington District of Columbia, Maryland, Virginia (CEAL DMV), is a multi-community and multi-university consortium. Through collaboration and shared leadership, the CEAL-DMV the consortium- comprising five institutions: George Washington University, Howard University, Johns Hopkins University, Morgan State University, and the University of Maryland, Baltimore-has established a regional structure for bi-directional community involvement to engender trust and foster communication. Each site builds on thriving community partnerships, which have been instrumental in enhancing trust, community capacity, and readiness to reduce health disparities.

DETAILED DESCRIPTION:
The investigators propose to evaluate the effect of a multi-level, community-digital health promotion intervention, compared to delayed control intervention, at improving health and social service utilization, and the prevention and management of hypertension, diabetes, overweight and obesity. The evidence-based intervention is based on substantial evidence supporting the role of Community Health Workers in health promotion and reduction of risks associated with chronic diseases.

Studies have demonstrated community health worker (CHW) intervention success at improving chronic disease risks and management, including for hypertension and diabetes, through support in implementing clinical recommendations, overcoming barriers to lifestyle behavior change, achieving personal goals, and preventing complications. Additionally, there is substantial evidence supporting digital approaches for the prevention and management of cardiometabolic diseases. The proposed intervention and methods also build on almost three years of CEAL DMV collaboration with community partners. At the community level, core activities will focus on capacity building to ensure the trusted community-based organization partners are fully supported in the implementation of community-digital strategies to address hypertension, diabetes, overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Black or Latino
* Age 18 years or older
* Reside in defined geographic area
* Diagnosis of one or more target conditions: Prediabetes/Diabetes (HbA1c 5.7%), Hypertension (≥130/80 mm Hg), Overweight/obesity (BMI >25 kg/m^2)

Exclusion Criteria:

* Unable to provide informed consent
* No access to phone/internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 664 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Service utilization as assessed by the number of participants who use referral services | 6 and 9 months
  Utilization will be calculated by the total number of participants who use services referred to by the community health workers.

SECONDARY OUTCOMES:
Satisfaction with health and health-related social services as assessed by a 3-point Likert Scale | 6 and 9 months
  Participants who utilize health and/or social services will be asked if satisfied with services received from health workers (i.e health care providers, mental health professionals and community health workers) using a a 3 point likert scale ranging from 1-3. Higher values would imply higher satisfaction).
Body mass index (BMI) in kg/m^2 | 6 and 9 months
  Body mass index (BMI) in kg/m^2 as assessed by weight-to-height ratio
Blood pressure | 6 and 9 months
  Systolic and diastolic blood pressure (mmHg)
Hemoglobin A1c (HbA1c) levels | 6 and 9 months
  Pre-diabetes and diabetes management as assessed by Hemoglobin A1c levels
Trust in health research and information sources as assessed by the Trust in Medical Research Survey | 6 and 9 months.
  Trust in Medical Research Survey, distrust sub-scale ranges from 0 to 20 with lower scores indicating better trust; trust sub-scale ranges from 0 to 24, higher scores mean better trust
Social determinants of health as assessed by the Health Related Social Needs Tool | 6 and 9 months.
  Health Related Social Needs Tool, scores ranging from 0 to 36; higher scored indicate higher need
Self-reported exercise frequency | 6 and 9 months
  Exercise frequency will be assessed by number of days per week a participant engages in moderate to strenuous exercise
Self-reported intake of regular soda or pop that contains sugar. | 6 and 9 months
  Participants will report the frequency of consumption of regular soda or pop that contains sugar each week. Higher number of times/week represents a worse outcome.
Self-reported sweetened fruit drinks intake | 6 and 9 months
  Participants will report the number of times they consumed sweetened fruit drinks per week. Higher number of times/week represents a worse outcome.
Self-reported fruit intake | 6 and 9 months
  Participants will report the frequency of consumption of fruits per week. Higher number of times/week represents a better outcome.
Self-reported intake of green leafy or lettuce salad | 6 and 9 months
  Participants will report the frequency of consumption of green leafy or lettuce salad each week. Higher number of number of times/week represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Himmelfarb, PhD, MSN, BS, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - George Washington University, Milken Institute of Public Health, Washington D.C., District of Columbia
  - Johns Hopkins University School of Nursing, Baltimore, Maryland